CLINICAL TRIAL: NCT06682689
Title: Integrative Investigation of Transcutaneous Vagus Nerve Stimulation: Impact on Postpartum Mental Health Through Wearable Technology, Hormonal Analysis and Modulatory Factors
Brief Title: Investigation of TVNS Administration on Postpartum Mental Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: German Center for Mental Health (DZPG) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: TUE/858/2023BO2
Record Dates: First submitted 2024-11-06; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-09

CONDITIONS: Postpartum Depression (PPD); Postpartum Anxiety; Postpartum Sadness; Postpartum Blues
Keywords: tVNS; Transcutaneous vagus nerve stimulation; Postpartum; PPD; Depression
MeSH Terms: conditions — Depression, Postpartum; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- High-low tVNS (Experimental): Participants in this group will be instructed to use the tVNS device every day for the first six weeks according to the manufacturer's guidelines, at an intensity where they can feel a tingling sensation but below the pain threshold. After six weeks (T2) of intervention, they will be asked to switch to a different protocol for the next six weeks, using the device at the lowest possible intensity. Additional instructions will be provided, and they will be informed that this stimulation uses different parameters set by the research team.
  Interventions: Device: transcutaneous vagus nerve stimulation
- Low-high tVNS (Active Comparator): Participants in this group will receive the inverted intervention, with the first six weeks of stimulation at the lowest possible intensity (0.1 mA) with the same instructions regarding duration of stimulations, followed by six weeks of high-intensity stimulation as instructed by the manufacturer.
  Interventions: Device: transcutaneous vagus nerve stimulation
- No tVNS (No Intervention): This group of participants will be included in all measurements (T1-T3) and check-ups, except for the tVNS stimulation.

INTERVENTIONS:
Device: transcutaneous vagus nerve stimulation — Two groups will use a tVNS stimulator for 12 weeks. Group 1 will apply active stimulation for up to 4 hours daily at a comfortable level for 6 weeks, while Group 2 will use it at the lowest intensity (0.1 mA). After 6 weeks (T2), the groups will switch. Participants will be instructed to use the device for at least 1 hour a day, with a recommendation of 4 hours, following guidelines and recent studies. The CE-certified tVNS® E device non-invasively stimulates the vagus nerve via the ear. It is approved for treating a.o.depression. Device parameters (intensity, pulse length, frequency) mimic invasive VNS techniques, ensuring safe and effective signal transmission. Stimulation will be applied to the left ear, with intensity adjusted to a tingling sensation, avoiding discomfort. The study follows an approved protocol, with low-intensity stimulation as a control. The device delivers biphasic impulses at 25 Hz, with 28 seconds ON and 32 seconds OFF, and is safe for extended use.
  Arms: High-low tVNS; Low-high tVNS

SUMMARY:
The aim of the study is to explore whether transcutaneous vagus nerve stimulation (tVNS) may be effective in preventing mood swings and depressive symptoms in the postpartum phase, as well as serving as a supplementary intervention in cases where mood symptoms develop. The study will investigate the effects of tVNS intervention during the first 12 weeks postpartum. Pregnant women will be recruited for the study, and the intervention will begin shortly after giving birth. Participants will receive different instructions on how to use the tVNS device. Additional parameters such as physiological functions, chronic stress, hormones, environment, and personality traits will also be assessed.

DETAILED DESCRIPTION:
The study uses a crossover, repeated-measures, within-subject, and between-subject placebo and active control design. Three groups of women who have recently given birth will receive either high-intensity tVNS, low-intensity tVNS, or no stimulation intervention for six weeks. After this period, the two tVNS groups will switch protocols for another six weeks. Participants will also undergo a battery of psychometric and neuropsychological tests at multiple time points. By applying a multilevel approach, the investigators will assess changes in postpartum mood and mental state from subjective (daily mood assessments, psychometric tests), cognitive (neuropsychological tests), physiological (heart rate, sleep patterns), and endocrine (cortisol, sex hormones) perspectives.

Throughout the study, all participants will answer app-based ecological momentary assessments (EMA) to monitor mood fluctuations after stimulation and compare outcomes. Participants' partners will be invited to take part in the study if they wish; they will complete questionnaires regarding their mental health and the perceived support they provide. During the initial screening, participants will receive detailed information about the study, and inclusion and exclusion criteria will be evaluated.

At the first meeting (T1), informed broad consent will be obtained, and the study will be explained in detail. Instructions for using the tVNS devices will be provided based on group assignments. Participants will complete questionnaires, undergo a short neuropsychological test, and provide hair samples for cortisol concentration analysis.

After giving birth, participants (or their partners, with permission) will notify the researchers, and each woman in the experimental tVNS groups will receive a package containing the stimulator and access to usage tutorials and instructions. All participants will also receive smartwatches with usage instructions.

The main study will include 120 women who have recently given birth, randomly assigned to one of three groups:

Group one (High-low tVNS) will first receive an active, high-intensity tVNS stimulation protocol for six weeks at a self-chosen level below the pain threshold and will be advised to use it for up to four hours a day (as per the device manual's full and maximal stimulation session). Precise instructions and protocols to assess the stimulation intensity will be given beforehand. After six weeks (T2), they will switch to the low-intensity tVNS protocol used by group two.

Group two (Low-high tVNS) will use the device at the lowest possible intensity of 0,1 milliampere. This intensity equals the intensity of stimulation during the "OFF" Phase, for more details see "Arms and interventions"". After six weeks, participants will switch protocol for the one provided at the begging for group one for the remaining six weeks.

The device is pre-programmed to stimulate with constant parameters (except for intensity), and to minimize placebo effects, participants will be informed that different protocols with varying sensations are being tested.

Group three (No stimulation) will not receive any tVNS stimulation. Their mood and symptoms will be assessed similarly to the other two groups, and physiological measures will be monitored via smartwatch and hair sampling.

At week six (T2; around the 6th-7th week postpartum), participants from all groups will visit the lab to complete questionnaires, provide hormone samples, and undergo neuropsychological assessments.

During the experimental phase, participants will report daily on their current mood. They will continue to complete repeated questionnaires assessing their mental health, quality of life, sleep quality, and symptoms of depression and anxiety. At two postpartum time points (T2 and T3; weeks 6 and 12 after parturition), participants will be asked to return for additional sessions where blood will be drawn for hormonal analysis, questionnaires will be repeated, and neuropsychological testing will be performed. At week 12, hair samples will again be collected for cortisol concentration analysis.

A voluntary online follow-up is planned after the study. At 6 and 9 months postpartum, participants will be invited to complete some of the standardised questionnaires, previously administered earlier in the study. These questionnaires will assess various aspects of their current state, including mental health, physical well-being, and parenting stress

The study utilizes the CE-certified tVNS® E device to non-invasively stimulate the vagus nerve, in compliance with European safety and performance standards (Class IIa, based on (EU) 2017/745 for medical devices, classified as a short-term, active therapeutic, non-invasive medical device under rule 9). This device stimulates the vagus nerve non-surgically by targeting the auricular branch of the vagus nerve, which interfaces with the skin at the cymba conchae of the external ear. The tVNS® E is approved for use in healthy participants, as well as for the following conditions (without restrictions for healthy participants, provided tVNS exclusion criteria are followed): treatment of seizures in pharmaco-resistant epilepsy with focal and/or generalized seizures (to reduce seizure frequency); adjunctive treatment of depression; treatment of emotional outbursts in Prader-Willi syndrome (to reduce frequency); adjunctive treatment of chronic migraine (to reduce headache frequency); and prophylactic migraine therapy for patients with chronic migraines who refuse or do not tolerate prophylactic medication (tVNS® E Instruction for Use, Version 1.6, 2023-01-30).

ELIGIBILITY:
Inclusion Criteria:

* No malformation of fetal organs (no abnormalities detected during "organ screening").
* Ability to provide written consent for themselves.
* Sufficient German language skills to communicate and understand study procedures.

Exclusion Criteria:

* Exclusion criteria for tVNS use (i.e., pregnancy, active implants such as cochlear implants or cardiac pacemakers, cerebral shunts, skin problems, cardiovascular health issues).
* Cardiac arrhythmias or coronary heart disease.
* Neurological disorders.
* Current diagnosis or episode of a mood disorder.
* Diagnosed schizophrenia spectrum and other psychotic disorders.
* Severe substance use disorders.
* Individual exclusion may also occur based on other health issues if the study clinician determines that participation in the study may pose a disadvantage for the participant or the child.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
tVNS-induced changes in postpartum depression symptoms | Measured during pregnancy (T1), 6 weeks after birth (T2), and 12 weeks after birth (T3)]
  To evaluate the effect of transcutaneous vagus nerve stimulation (tVNS) on depressive symptoms, as measured by the Edinburgh Postpartum Depression Scale (EPDS), which ranges from 0 to 30, with higher scores indicating more severe depressive symptoms. A standard cut-off score of 12-13 is typically used to indicate probable depressive symptoms. The total EPDS score will be assessed at multiple time points throughout the study, allowing for the comparison of changes in depressive symptom trajectories across conditions (tVNS vs. control). This design aims to capture differences in the development and progression of depressive symptoms between groups over the course of pregnancy and postpartum.
tVNS-induced changes in the daily mood | From the recruitment through first 12 weeks of postpartum period
  The study will track and analyze the daily trajectory of mood changes-both positive and negative-from a baseline period prior to the 6-week transcutaneous vagus nerve stimulation (tVNS) intervention and throughout the intervention period, with assessments concluding on the final day of the intervention. Daily mood changes and stability will be measured using the Positive and Negative Affect Schedule (PANAS), administered through app-based ecological momentary assessment (EMA). Each item on the PANAS is rated on a 5-point Likert scale, ranging from 1 ("gar nichts" / "not at all") to 5 ("äußerst" / "extremely"), with higher scores reflecting a greater intensity of the specified mood. Positive affect (PA) scores represent more positive mood states (higher scores indicating better mood), while negative affect (NA) scores indicate the severity of negative mood states (higher scores representing worse mood).
  The analysis will focus on identifying trends, patterns, and fluctuations in mood

SECONDARY OUTCOMES:
Intervention acceptance analysis | through study completion, an average of 6 months
  Using a mixed-method approach, including compliance analysis (tracking the frequency and duration of tVNS device use), retention analysis (comparing retention and dropout rates between groups at different time points), and post-intervention questionnaire-based data on participants' satisfaction with the intervention (assessing the burden of the intervention, side effects, and participants' theoretical willingness to recommend it to others).
Heart-rate variability changes | From the recruitment through first 12 weeks of postpartum period
  HRV will be assessed through smartwatches, with analyses focusing on tVNS-induced changes compared to controls using RMSSD (Root Mean Square of Successive Differences), SDNN (Standard Deviation of NN intervals), and frequency-domain methods.
Subjective sleep quality changes | through study completion, an average of 6 months
  Subjective sleep quality will be assessed monthly using the Pittsburgh Sleep Quality Index (PSQI), along with an ecological momentary assessment (EMA) question about sleep quality. Group comparisons will determine whether tVNS induces changes in sleep quality compared to control conditions.
  In scoring the PSQI, seven component scores are derived, each rated from 0 (no impairment) to 3 (severe impairment). The component scores are summed to produce a global score (range 0 to 21), with higher scores indicating poorer sleep quality.
Objective sleep quality | through study completion, an average of 6 months
  Sleep quality (duration, depth, and regularity) will be measured objectively using smartwatch data, focusing on tVNS-induced changes compared to the control group. Sleep duration will be measured in hours and minutes, sleep depth will be assessed based on time spent in different sleep stages (light sleep, deep sleep, and REM) in minutes, and sleep regularity will be evaluated by the variability in sleep and wake times, also in hours and minutes. Those submeasures will be further analysed to an overall sleep quality outcome
  Note: While smartwatches provide estimates, their limitations in accuracy are acknowledged, and subjective data will be triangulated with these measures.
Postpartum depression diagnosis (clinical threshold) | From the birth of the child to the end of the study (12 weeks)
  The number of women in each group who develop clinical threshold scores on the EPDS will be compared to assess whether tVNS reduces the risk of postpartum depression compared to controls.
Objective measure of chronic stress | Two measurements: During pregnancy (T1) and 12 weeks postpartum (T3)
  Hair cortisol concentrations will be measured twice (T1 during pregnancy, and T3 at 12 weeks postpartum) to assess tVNS-induced changes in chronic stress levels from past three months compared to controls. Individual events causing massive changes in cortisol concentration will be noted.
Subjective chronic stress levels | Three times: During 1st visit, at 6 weeks postpartum and 12 weeks after birth
  Total score on the Trier inventory for chronic stress (TICS; Schulz et al., 2004)
Daily activity changes induced by tVNS | From the recruitment through first 12 weeks of postpartum period
  Daily activity will be measured via smartwatch data, focusing on activity level changes between the tVNS and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Derntl, Prof., PhD, Principal Investigator — University Hospital Tübingen; Nils Kroemer, Prof., Dr. rer. nat., Principal Investigator — University Hospital Tübingen
Locations (1):
- University Hospital Tuebingen; Department of Psychiatry and Psychotherapy, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) will be anonymized and shared in accordance with the GDPR. Data will be shared to the extent that re-identification is not possible.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be open to access after the analysis and publication by the study officials.
Access Criteria: The protocols, plans, and codes and IPD will be shared via open-access platforms and linked to the publication. Specific data not available online will be provided upon request by one of the corresponding authors.